CLINICAL TRIAL: NCT06138964
Title: Randomized Intra-individually Controlled Double-blinded Trial Comparing Effect of Small Interfering RNA Against SPARC (siSPARC) Microneedle Patch Versus Small Interfering RNA Against SPARC and IL4-RA (siSPARC + siLR4A) Microneedle Patch on Appearance of Post-surgical Scars
Brief Title: Comparing the Effect of siSPARC Microneedle Patch Versus siSPARC+siLR4A Microneedle Patch on Post-surgical Scars
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Skin Centre (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022/00942
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Keloid; Wound Heal; Wound
MeSH Terms: conditions — Keloid; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- siSPARC microneedle patch (Experimental): siSPARC microneedle patch
  Interventions: Drug: siSPARC microneedle patch
- siSPARC + siLR4A microneedle patch (Experimental): siSPARC + siLR4A microneedle patch
  Interventions: Drug: siSPARC + siLR4A microneedle patches

INTERVENTIONS:
Drug: siSPARC + siLR4A microneedle patches — siSPARC + siLR4A microneedle patch
  Other Names: siSPARC + siLR4A microneedle patch
  Arms: siSPARC + siLR4A microneedle patch
Drug: siSPARC microneedle patch — siSPARC microneedle patch
  Other Names: siSPARC + siLR4A microneedle patch
  Arms: siSPARC microneedle patch

SUMMARY:
This randomized, double-blind controlled study aims to compare the effect on appearance of post- surgical scars between daily application of siSPARC microneedle patch versus siSPARC + siLR4A microneedle patches. These are patches comprising short microneedles embedded with hydrolysed RNA (siRNAs).

DETAILED DESCRIPTION:
This is an 8-week, single centre double-blinded intra-individually controlled trial to compare the effect of daily application of siSPARC microneedle patch versus siSPARC + siLR4A microneedle patch on post-surgical scars. At least 50 subjects will be recruited for the study. After the patients have been screened for study eligibility by the study investigators or coordinators, the subjects who have understood and signed the informed consent will be enrolled in the study. Provided a subject satisfies all inclusion criteria and does not fall within exclusion criteria during the screening visit, that subject will be started on the trial during that same visit. Computer-generated randomisation will be performed to determine the randomization of patient population to the siSPARC microneedle patch or siSPARC + siLR4A microneedle patch. Subsequent follow-up visits would be on Day 30 and Day 60. A deviation of +/- 7 days will be accepted during the follow-up. Each study visit will last between 30-60 minutes.

Study investigators and coordinators will be performing the following assessments:

1. High resolution 3D imaging: Scar elevation will be measured using the Space Spider 3D scanner, with a resolution of 0.1 mm and a blue light-emitting diode (LED) light source;
2. Vancouver scar scale (VSS) score;
3. Scar Cosmesis Assessment and Rating (SCAR) scale score from the photographs;
4. Change in patient-reported levels of pain and itch using a 11-point numerical rating scale; and
5. Assessment of side effects (if any). Photographic documentation: Photographic documentation will be performed at baseline and during the specified follow-up examinations. Images will be taken with standardized camera settings and standardized positioning of the subject. These images will be assessed by investigators to assess the change in scar appearance.

The siRNA microneedle patches are not commercially available. These patches have undergone testing with guinea pigs and white rabbits and were ascertained as a 'non-sensitiser' and 'non- irritant', respectively. The patches have also underwent testing to L-929 cells which are adherent cells of mouse fibroblast cell line and found to be 'non-cytotoxic'. This study involves a trial comparing treatment outcomes; there is no investigative work conducted and hence no incidental findings are not anticipated.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Age 21-75
* 2 weeks (+/- 7 days) after surgical operation with incision into the dermis
* Post-stitch removal when stitches were applied
* Wound closure/union achieved

Exclusion Criteria:

* Pregnant or lactating participant
* Participants with wound infection
* Participants assessed to be uncooperative or unable to self-administer the interventions
* Participants with known contact allergy to ingredients in the patch formulation (comprising hyaluronic acid, siRNA and glue) and/or isopropyl alcohol
* Participants who are unable to personally consent (for e.g., cognitively impaired)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-11-14 (Estimated); Study Completion 2024-11-14 (Estimated)

PRIMARY OUTCOMES:
Assessment of post-surgical scar elevation | 1 year
  To compare the efficacy in reducing post-surgical scar elevation between daily application of siSPARC microneedle patch versus siSPARC + siLR4A microneedle patch. This will be measured using high resolution 3D imaging: scar elevation will be measured using the Space Spider 3D scanner, with a resolution of 0.1 mm and a blue LED light source. The lower the elevation, the better the outcome.

SECONDARY OUTCOMES:
Assessment of Vancouver Scar Scale (VSS) score | 1 year
  To evaluate the differences in VSS scores between daily application of siSPARC microneedle patch or siSPARC + siLR4A microneedle patch. The total VSS score is based on 4 points: (1) vascularity (on a scale of 0 being normal to 3 being purple); (2) pigmentation (on a scale of 0 being normal, to 2 being hyperpigmentation); (3) pliability (on a scale of 0 being normal to 5 being contractures); and (4) height (on a scale of normal being flat to 3 being >5mm). Higher scores indicate a worse outcome.
Assessment of Scar Cosmesis Assessment and Rating (SCAR) Scale | 1 year
  Assessment of SCAR Scale performed on photographs. The SCAR Scale is based on 8 points: (1) scar spread (on a scale of 0 being none to near-invisible to 4 being severe); (2) erythema (on a scale of 0 being none to 3 being deep red or purple); (3) dyspigmentation (being either 0 absent or 1 present); (4) track or suture marks (being either 0 absent or 1 present); (5) hypertrophy or atrophy (on a scale of 0 being none to 3 being severe); (6) impression (being either 0 desirable or 1 undesirable); (7) patient reported itch in last 24 hours (being either 0 absent or 1 present); and (8) patient reported pain (being either 0 absent or 1 present). Higher scores indicate a worse outcome.
Patient-reported levels of pain and itch using a 11-point numerical rating scale | 1 year
  Patient-reported levels of pain and itch using a 11-point numerical rating scale from 0 to 10 (0 being no pain, and 10 being the worst pain). Higher scores indicate a worse outcome.
Side effects | 1 year
  Patient reported side effects (if any), such as contact dermatitis (if any).

CONTACTS AND LOCATIONS:
Overall Officials: Hong Liang Tey, Principal Investigator — National Skin Centre
Locations (1):
- National Skin Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No